CLINICAL TRIAL: NCT03750279
Title: Inflammatory Targeted Low-level Laser Treatment of Knee Osteoarthritis - A Randomized Clinical Trial
Brief Title: Inflammatory Targeted Laser Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bergen KOA laser RCT
Record Dates: First submitted 2018-11-06; First posted 2018-11-23 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Inflammation; Photobiomodulation; Low-level laser therapy; Double-blind; Randomized clinical trial; RCT
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation | interventions — Exercise Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two laser devices of the same appearance are used, i.e. one with 3x60 mW output power and one with 0 mW output power (sham). Participants in one group is treated with the sham laser device and the other group is treated with laser. The laser beam is invisible for the eye (wavelength 904 nm) and of such low power that heat is not detected. Thus, the participants, therapists and assessors are unaware of which laser device is active/inactive. The laser devices were randomly coded by a secretary who is not otherwise involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise therapy + LLLT (Active Comparator): * Exercise therapy 3 times per week for 8 weeks from baseline.
  * LLLT applied to the knee 3 times per week for 3 weeks from baseline.
  Interventions: Other: Exercise therapy; Other: LLLT
- Exercise therapy + sham LLLT (Placebo Comparator): * Exercise therapy 3 times per week for 8 weeks from baseline.
  * Sham LLLT applied to the knee 3 times per week for 3 weeks from baseline.
  Interventions: Other: Exercise therapy; Other: Sham LLLT

INTERVENTIONS:
Other: Exercise therapy — * 5 min. warm up with light exercises for the lower limb prior to strength/endurance exercise therapy.
  * Strength/endurance exercise therapy including level 1 or 2 per session:
  Level 1: Pelvic lifts (2x15 rep.), one-legged knee bends (2x10 rep. per leg), hip abductions (2x10 rep. per leg). The participants may progress from level 1 to level 2.
  Level 2: Pelvic lifts (3x15 rep.), one-legged knee bends (3x10 rep. per leg), hip abductions (2x10 rep. per leg), sideways slide (2x10 rep. per leg), and backwards slide (2x10 rep. per leg). The participants may regress from level 2 to level 1.
Other: LLLT — - LLLT (60 mW mean output per probe, 904 nm wavelength) applied to the knee in adherence with the recommendations by World Association for Laser Therapy, in terms of dosage per treatment spot.
  Arms: Exercise therapy + LLLT
Other: Sham LLLT — - Same procedure as in the LLLT group with the exception of laser irradiation (0 mW mean output power).
  Arms: Exercise therapy + sham LLLT

SUMMARY:
This study is conducted to evaluate the effectiveness of low-level laser therapy (LLLT) as an adjunct to exercise therapy in knee osteoarthritis (KOA).

ELIGIBILITY:
Inclusion criteria:

* Any gender
* Age ≥ 50 years
* Pain on movement ≥ 40 mm Visual Analog Scale
* Knee pain for the last ≥ 3 months
* KOA verified with the American College of Rheumatology criteria using a history and physical examination, i.e. knee pain and at least three of the following: ≥ 50 years old, ≤ 30 minutes of morning stiffness, crepitus on active range of motion, bony tenderness, bony enlargement, and no palpable warmth of synovia

Exclusion criteria:

* Knee alloplastic
* Total meniscectomy
* Intra-articular steroid injection and/or oral steroid treatment within the last six months
* Cancer
* Rheumatoid arthritis
* Severe cognitive deficit
* Neurological deficits affecting the knee
* Inability to speak and understand English/Norwegian

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Pain on movement | 0, 3, 8, 26 and 52 weeks after randomization
  The participants are asked to rate their pain experienced on movement using an unidimensional visual analogue scale (VAS). "No pain" (0) is written in one end and "worst imaginable pain" (100) is written in the other end of the VAS tool.
Pain at night | 0, 3, 8, 26 and 52 weeks after randomization
  The participants are asked to rate their pain experienced in bed at night using an unidimensional visual analogue scale (VAS). "No pain" (0) is written in one end and "worst imaginable pain" (100) is written in the other end of the VAS tool.
Pain at rest | 0, 3, 8, 26 and 52 weeks after randomization
  The participants are asked to rate their pain experienced at rest in sitting position using an unidimensional visual analogue scale (VAS). "No pain" (0) is written in one end and "worst imaginable pain" (100) is written in the other end of the VAS tool.
Pain in general | 0, 3, 8, 26 and 52 weeks after randomization
  Pain in general is reported with the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire pain subscale. The subscale is based on Likert scales, each with five severity categories. The raw KOOS score is transformed to a 0-100 percentage score (higher is better).

SECONDARY OUTCOMES:
Physical function in daily living | 0, 3, 8, 26 and 52 weeks after randomization
  Physical function in daily living is reported with the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire physical function in daily living subscale. The subscale is based on Likert scales, each with five severity categories. The raw KOOS score is transformed to a 0-100 percentage score (higher is better).
Physical function in sports and recreational activities | 0, 3, 8, 26 and 52 weeks after randomization
  Physical function in sports and recreational activities is reported with the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire physical function in sports and recreational activities subscale. The subscale is based on Likert scales, each with five severity categories. The raw KOOS score is transformed to a 0-100 percentage score (higher is better).
Quality of life | 0, 3, 8, 26 and 52 weeks after randomization
  Quality of life is reported with the Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire quality of life subscale. The subscale is based on Likert scales, each with five severity categories. The raw KOOS score is transformed to a 0-100 percentage score (higher is better).
Global health status assessment | 8 weeks after randomization
  The participants evaluate their change from baseline in terms of symptoms in general from 1 to 7 (1, no symptoms; 7, worse than ever).
Real time ultrasonography assessment of effusion | 0, 3, 8, 26 and 52 weeks after randomization
  Maximum height will be measured.
Real time ultrasonography assessment of neovascularization | 0, 3, 8, 26 and 52 weeks after randomization
  Doppler area will be measured.
Real time ultrasonography assessment of femur cartilage thickness | 0, 3, 8, 26 and 52 weeks after randomization
30 seconds chair stand | 0, 3, 8, 26 and 52 weeks after randomization
  Last attempt counts if the participant is more than half way up.
Knee extension active range of motion | 0, 3, 8, 26 and 52 weeks after randomization
  A 30 cm goniometer is used.
Knee flexion active range of motion | 0, 3, 8, 26 and 52 weeks after randomization
  A 30 cm goniometer is used.
Maximum pain free isometric quadriceps strength | 0, 3, 8, 26 and 52 weeks after randomization
  A dynamometer is used: The dynamometer display is not visible during the procedure in order to blind the assessor for the level of pressure.
Joint line pain pressure threshold | 0, 3, 8, 26 and 52 weeks after randomization
  The most tender spot in the medial knee joint line is identified with palpation. Subsequently, a pain pressure threshold algometer is used at this spot. The display of the algometer is not visible during the procedure in order to blind the assessor for the level of pressure.
Tibia bone pain pressure threshold | 0, 3, 8, 26 and 52 weeks after randomization
  The most tender spot in the medial knee joint line is identified with palpation. Subsequently, a pain pressure threshold algometer is used 1.5 cm distally from this spot. The display of the algometer is not visible during the procedure in order to blind the assessor for the level of pressure.
Analgesic drug consumption due to knee pain | 0, 3, 8, 26 and 52 weeks after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No